CLINICAL TRIAL: NCT00860509
Title: Phyteaux-II- Regulation of Cholesterol Absorption: Response of LDL to Low and Naturally High Phytosterol Diets
Brief Title: Comparison of Low and High Phytosterol Diets With Respect to Cholesterol Metabolism
Acronym: Phyteaux-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Richard Ostlund/Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PBRC26030
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease
Keywords: phytosterols; cholesterol excretion; cholesterol absorption; diet; mass spectrometry; deuterium
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Phytosterol Diet (Placebo Comparator): Diet with 100 mg of daily phytosterols
  Interventions: Other: Low Phytosterol and High Phytosterol Diets
- High Phytosterol Diet (Active Comparator): Diet with 600 mg of daily phytosterols
  Interventions: Other: Low Phytosterol and High Phytosterol Diets

INTERVENTIONS:
Other: Low Phytosterol and High Phytosterol Diets — Diets with 600 or 100 mg of daily phytosterols for 4 weeks were given to each subject, in random order

SUMMARY:
The objective of this study is to compare cholesterol absorption and metabolism after feeding diets naturally low or high in phytosterols. All meals will be prepared in a metabolic kitchen and analyzed for phytosterols. In a randomized crossover design a group of up to 25 healthy subjects will consume diets containing either 100 mg/day or 600 mg/day phytosterols for 4 weeks. At the end of each dietary period percent cholesterol absorption, fecal cholesterol excretion and LDL cholesterol level will be measured. The hypothesis is that LDL cholesterol and cholesterol excretion will be improved on the high phytosterol diet even though macronutrient composition, mineral intake and fiber consumption are similar.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race or ethnicity between 18 to 80 years of age, inclusive;
* Body mass index between 20-35 kg/m2;
* LDL-cholesterol between 100-189 mg/dL based on the average of duplicate screening measures. If the two LDL-C levels differ by more than 30 mg/dL, a third test will be scheduled with all three results averaged;
* Free of chronic disease;
* Willing to eat only the foods that are provided by the Center during the diet periods;
* Willing to consume no more than 1 alcoholic drink per day.
* Willing to abstain from the consumption of alcohol for 48-hours prior to blood draw days;
* Willing to drink no more than 5 cups of caffeine-containing beverages a day.

Exclusion Criteria:

* Age < 18 or > 80 years;
* Based on duplicate screening laboratory values: 1) LDL-C > or = 190 mg/dL; 2) TG > or = 250 mg/dL; 3) blood pressure > or = 160 mm Hg systolic or 95 mm Hg diastolic;
* Documented presence of atherosclerotic disease;
* Diabetes mellitus;
* Renal, hepatic, endocrine, gastrointestinal, hematological or other systemic disease;
* Body mass index > 35;
* For women, pregnancy, breast feeding or postpartum < 6 months;
* For women, peri-menopausal;
* History of drug or alcohol abuse;
* History of depression or mental illness requiring treatment or medication within the last 6 months;
* Multiple food allergies or significant food preferences or restrictions that would interfere with diet adherence;
* Chronic use of over-the-counter medication which would interfere with study endpoints including laxatives and antacids;
* Lifestyle or schedule incompatible with the study protocol;
* Planned continued use of dietary supplements through the study trial;
* Taking any lipid-lowering, or other medications known to affect blood cholesterol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Fecal cholesterol excretion | At the end of week 4 on each diet

SECONDARY OUTCOMES:
Intestinal cholesterol absorption | At the end of week 4 on each diet

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ostlund, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Pennington Biomedical Research Center-Louisana State University System, Baton Rouge, Louisiana, United States

REFERENCES:
- [Result] Lin X, Racette SB, Lefevre M, Spearie CA, Most M, Ma L, Ostlund RE Jr. The effects of phytosterols present in natural food matrices on cholesterol metabolism and LDL-cholesterol: a controlled feeding trial. Eur J Clin Nutr. 2010 Dec;64(12):1481-7. doi: 10.1038/ejcn.2010.180. Epub 2010 Sep 1. PMID 20808333